CLINICAL TRIAL: NCT03901456
Title: Care to Plan: Preliminary Efficacy of a Tailored Resource for Family Members of Persons With Dementia
Brief Title: Care to Plan: a Tailored Resource for Family Members of Persons With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00005971; 1R21AG060419-01A1 (NIH)
Record Dates: First submitted 2019-03-28; First posted 2019-04-03 (Actual); Results first posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-06

CONDITIONS: Dementia; Alzheimer Disease; Memory Loss
Keywords: Caregiving
MeSH Terms: conditions — Dementia; Alzheimer Disease; Memory Disorders

STUDY DESIGN:
Intervention Model Description: Phase I of the study will include enrollment of 20 participants to test and refine the online tool [non-randomized]; in Phase II, we aim to enroll 100 participants to generate preliminary evaluation data [randomized].
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase II [Randomized]: Treatment (Experimental): Participants randomized to this treatment arm will receive the Care to Plan (CtP) intervention as a part of Phase II.
  Interventions: Behavioral: Care to Plan
- Phase II [Randomized]: Control (Active Comparator): Participants randomized to a usual care control group as a part of Phase II.
  Note: If eligible, participants in this control group will be asked if they are interested in enrolling in a similar, additional feature of the study to test the Care to Plan tool following the initial 6-month study.
  Interventions: Behavioral: Usual Care
- Phase I [Non-randomized]: Treatment (Experimental): Participants enrolled in Phase I of the project to receive the intervention [non-randomized; no comparison group].
  Interventions: Behavioral: Care to Plan

INTERVENTIONS:
Behavioral: Care to Plan — Care to Plan (CtP) is an online care planning tool that provides a succinct and clear overview of various types of ADRD caregiver interventions, administers a brief validated assessment of risk, and generates individualized service recommendations for Alzheimer's disease and related dementia (ADRD) caregivers as well as resources that link users to a selected recommendation. Caregivers will complete the tool with the guidance of a CtP interventionist (Senior Care Navigator/Riverside Health System staff). The interventionist will discuss CtP recommendations with caregivers and help caregivers enroll in a recommended support service if so desired.
  Arms: Phase I [Non-randomized]: Treatment; Phase II [Randomized]: Treatment
Behavioral: Usual Care — Receive care as usual.
  Note: If eligible, participants in this control group will be asked if they are interested in enrolling in a similar, additional feature of the study to test the Care to Plan tool following the initial 6-month study.
  Arms: Phase II [Randomized]: Control

SUMMARY:
The present study will refine and conduct a preliminary efficacy evaluation of Care to Plan. Care to Plan is an online care planning tool that provides a succinct and clear overview of various types of dementia caregiver interventions, administers a brief validated assessment of risk, and generates individualized recommendations for dementia caregivers as well as resources that link users to a selected recommendation.

There remains a lack of individualized information that can directly meet the diverse needs of caregivers or their relatives with Alzheimer's disease or a related dementia (ADRD). This project will advance scientific knowledge, technical capability, and clinical practice as they pertain to ADRD management and caregiver support.

DETAILED DESCRIPTION:
Given the well-documented health implications of dementia family caregiving, existing interventions are designed to modify the more challenging aspects of care for a relative with Alzheimer's disease or a related dementia (ADRD) in order to improve key outcomes. However, current research has yet to discern which caregivers are most likely to benefit from different types of interventions or services. There also remains a lack of individualized information that can directly meet the heterogeneous needs of caregivers or their relatives with ADRD. This project will advance scientific knowledge, technical capability, and clinical practice as they pertain to ADRD management and caregiver support. The research team has developed and tested the feasibility and utility of an online care planning tool prototype (called Care to Plan, or CtP) that provides a succinct and clear overview of various types of ADRD caregiver interventions, administers a brief validated assessment of risk, and generates individualized service recommendations for ADRD caregivers as well as resources that link users to a selected recommendation. The goal of CtP is to offer a more efficient, user-directed process to link ADRD caregivers to the services that may be most appropriate for them given their needs, the needs of their relatives, and other contextual characteristics. We will deploy and more fully evaluate CtP for family caregivers of persons with ADRD who seek services in Riverside Health System (RHS) in the state of Virginia. The Specific Aims are to: 1) Implement CtP for 20 family members of persons with ADRD in four RHS clinical sites (Phase I) over a 1-month period; and 2) Evaluate the preliminary efficacy and implementation of CtP (Phase II) via an embedded randomized controlled evaluation for 100 newly enrolled ADRD caregivers over a 6-month period. We anticipate that the CtP will serve as an innovative, low-cost tool that both families and long-term service and support providers can utilize to better meet the diverse needs of family caregivers of persons with ADRD in their communities.

ELIGIBILITY:
Inclusion Criteria: The care recipient has received a provider diagnosis of Alzheimer's disease or a related dementia (ADRD); and 2) the caregiver is 21 years of age or older; 3) English-speaking; 4) self-identifies as someone who provides help to the person with ADRD because of their cognitive impairments; 5) the caregiver indicates a willingness to use Care to Plan (CtP); and 6) caregiver resides in one of 4 Riverside Health regions (based on zip code).

Exclusion Criteria: Those who do not meet the inclusion criteria above are not eligible. Additionally, those who endorse a history of a serious mental health disorder whose: a) symptoms have exacerbated in the last six months, and b) are not receiving steady, ongoing pharmacological or other treatment for these symptoms, will be excluded from the project.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph E Gaugler, PhD, Principal Investigator — University of Minnestoa
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
Public access to the research data generated from this project will be offered via de-identified data files maintained by the investigators. All personal identifiers of family caregivers of persons with Alzheimer's disease or a related dementia (ADRD) participating in the study will be removed and replaced with random identification numbers prior to distributing data files. Dr. Gaugler plans to maintain all data from the proposed project on the secure School of Public Health shared server folder for 7 years following study completion. Potential external investigators will be asked to complete a data use agreement and a recommended citation to these materials will be provided. Dr. Gaugler will oversee the distribution of public data during the course of the funding period and for an indefinite time thereafter.

REFERENCES:
- [Background] Pearlin LI, Mullan JT, Semple SJ, Skaff MM. Caregiving and the stress process: an overview of concepts and their measures. Gerontologist. 1990 Oct;30(5):583-94. doi: 10.1093/geront/30.5.583. PMID 2276631
- [Background] Fortinsky RH, Kercher K, Burant CJ. Measurement and correlates of family caregiver self-efficacy for managing dementia. Aging Ment Health. 2002 May;6(2):153-60. doi: 10.1080/13607860220126763. PMID 12028884
- [Background] Radloff, L. S. (1977). The CES-D Scale: A Self-Report Depression Scale for Research in the General Population. Applied Psychological Measurement, 1(3), 385-401. https://doi.org/10.1177/014662167700100306

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Sixty-five participants consented to participate (during Phase I or Phase II of the project). Two participants did withdrew or were lost to follow up prior to initial survey completion. Data is reported for 63 participants completing the initial survey.
Groups:
- Phase I: Treatment [Non-randomized]: Participants enrolled in Phase I of the project to receive the intervention [non-randomized, no comparison group].
  Care to Plan: Care to Plan (CtP) is an online care planning tool that provides succinct and clear overview of various types of ADRD caregiver interventions, administers a brief validated assessment of risk, and generates individualized service recommendations for Alzheimer's disease and related dementia (ADRD) caregivers as well as resources that link users to a selected recommendation. Caregivers will complete the tool with the guidance of a CtP interventionist (Senior Care Navigator/Riverside Health System staff). The interventionist will discuss CtP recommendations with caregivers and help caregivers enroll in a recommended support service if so desired.
- Phase II: Treatment [Randomized]: Participants in the treatment arm will receive the Care to Plan (CtP) intervention as part of Phase II.
  Care to Plan: Care to Plan (CtP) is an online care planning tool that provides a succinct and clear overview of various types of ADRD caregiver interventions, administers a brief validated assessment of risk, and generates individualized service recommendations for Alzheimer's disease and related dementia (ADRD) caregivers as well as resources that link users to a selected recommendation. Caregivers will complete the tool with the guidance of a CtP interventionist (Senior Care Navigator/Riverside Health System staff). The interventionist will discuss CtP recommendations with caregivers and help caregivers enroll in a recommended support service if so desired.
- Phase II: Control [Randomized]: Participants randomized to a usual care control group as part of Phase II.
  Note: If eligible, participants in this control group will be asked if they are interested in enrolling in a similar, additional feature of the study to test the Care to Plan tool following the initial 6-month study.
  Usual Care: Receive care as usual.
  Note: If eligible, participants in this control group will be asked if they are interested in enrolling in a similar, additional feature of the study to test the Care to Plan tool following the initial 6-month study.
Period: Overall Study
Arm/Group | Phase I: Treatment [Non-randomized] | Phase II: Treatment [Randomized] | Phase II: Control [Randomized]
Started | 20 | 22 | 21
Completed | 20 | 21 | 20
Not Completed | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment [Randomized]: Participants in the treatment arm will receive the Care to Plan (CtP) intervention as part of Phase II.
  Care to Plan: Care to Plan (CtP) is an online care planning tool that provides a succinct and clear overview of various types of ADRD caregiver interventions, administers a brief validated assessment of risk, and generates individualized service recommendations for Alzheimer's disease and related dementia (ADRD) caregivers as well as resources that link users to a selected recommendation. Caregivers will complete the tool with the guidance of a CtP interventionist (Senior Care Navigator/Riverside Health System staff). The interventionist will discuss CtP recommendations with caregivers and help caregivers enroll in a recommended support service if so desired.
- Control [Randomized]: Participants randomized to a usual care control group as part of Phase II.
  Note: If eligible, participants in this control group will be asked if they are interested in enrolling in a similar, additional feature of the study to test the Care to Plan tool following the initial 6-month study.
  Usual Care: Receive care as usual.
  Note: If eligible, participants in this control group will be asked if they are interested in enrolling in a similar, additional feature of the study to test the Care to Plan tool following the initial 6-month study.
- Total: Total of all reporting groups
Arm/Group | Treatment [Randomized] | Control [Randomized] | Phase I: Treatment [Non-randomized] | Total
Number analyzed (Participants) | 22 | 21 | 20 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.33 (16.54) | 63.38 (11.77) | 66.68 (11.43) | 63.24 (12.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 18 | 50
  Male | 5 | 6 | 2 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 22 | 21 | 20 | 63
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 4 | 5 | 12
  White | 18 | 17 | 15 | 50
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Caregiver Self-efficacy
Description: Eight-item survey developed by Fortinsky and colleagues. Responses for each item range from 1 (Very unconfident) to 5 (Very confident), with higher scores indicating greater self-efficacy. The 8-item responses are averaged. Mean of participant scores is reported.
Time Frame: Phase II Baseline, 3-months, 6-months
Population: Outcome reported for Phase II only; number analyzed varies by treatment arm and timepoint (due to missing data and/or withdrawal).
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Phase II [Randomized]: Treatment: Participants in the treatment arm will receive the Care to Plan (CtP) intervention as part of Phase II.
  Care to Plan: Care to Plan (CtP) is an online care planning tool that provides a succinct and clear overview of various types of ADRD caregiver interventions, administers a brief validated assessment of risk, and generates individualized service recommendations for Alzheimer's disease and related dementia (ADRD) caregivers as well as resources that link users to a selected recommendation. Caregivers will complete the tool with the guidance of a CtP interventionist (Senior Care Navigator/Riverside Health System staff). The interventionist will discuss CtP recommendations with caregivers and help caregivers enroll in a recommended support service if so desired.
- Phase II [Randomized]: Control: Participants randomized to a usual care control group as part of Phase II. Note: If eligible, participants in this control group will be asked if they are interested in enrolling in a similar, additional feature of the study to test the Care to Plan tool following the initial 6-month study.
  Usual Care: Receive care as usual. Note: If eligible, participants in this control group will be asked if they are interested in enrolling in a similar, additional feature of the study to test the Care to Plan tool following the initial 6-month study.
Arm/Group | Phase II [Randomized]: Treatment | Phase II [Randomized]: Control
Number analyzed (Participants) | 22 | 21
scores on a scale
  Baseline [Phase II] | 3.62 (.85) | 3.36 (.74)
  3-months [Phase II]: number analyzed (Participants) | 19 | 18
  3-months [Phase II] | 3.84 (.96) | 3.57 (.88)
  6-months [Phase II]: number analyzed (Participants) | 16 | 16
  6-months [Phase II] | 3.58 (.73) | 3.55 (.70)

2. Secondary Outcome: Care to Plan Service Use
Description: This author-developed scale is a self-report of a various services used over a 3 month period. Service types include Skills building, Problem solving, Take a break, Brain health, Support groups, Change your thinking, High powered combinations, and Other. The total number of services used are summed (ranging 0 to 8, with higher numbers indicating greater service use). The average of participant responses is reported.
Time Frame: Phase II Baseline, 3-months, 6-months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: services
Groups:
- Phase II[Randomized]: Treatment: Participants in the treatment arm will receive the Care to Plan (CtP) intervention as part of Phase II.
  Care to Plan: Care to Plan (CtP) is an online care planning tool that provides a succinct and clear overview of various types of ADRD caregiver interventions, administers a brief validated assessment of risk, and generates individualized service recommendations for Alzheimer's disease and related dementia (ADRD) caregivers as well as resources that link users to a selected recommendation. Caregivers will complete the tool with the guidance of a CtP interventionist (Senior Care Navigator/Riverside Health System staff). The interventionist will discuss CtP recommendations with caregivers and help caregivers enroll in a recommended support service if so desired.
Arm/Group | Phase II[Randomized]: Treatment | Phase II [Randomized]: Control
Number analyzed (Participants) | 22 | 21
services
  Baseline [Phase II] | 2.69 (1.25) | 2.62 (1.32)
  3-month [Phase II]: number analyzed (Participants) | 19 | 18
  3-month [Phase II] | 3.00 (0.88) | 2.56 (1.69)
  6-month [Phase II]: number analyzed (Participants) | 16 | 16
  6-month [Phase II] | 2.31 (1.20) | 2.25 (1.07)

3. Secondary Outcome: Phase II - Caregiver Distress: Role Overload
Description: A 3-item scale measuring caregivers' feelings of emotional fatigue. Item responses range from 1 = strongly disagree to 5 = strong agree. Item responses are averaged, with higher score representing greater role overload.
Time Frame: Phase II Baseline, 3-months, 6-months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale (mean)
Arm/Group | Phase II [Randomized]: Treatment | Phase II [Randomized]: Control
Number analyzed (Participants) | 22 | 21
score on a scale (mean)
  Baseline [Phase II] | 3.23 (1.28) | 3.71 (1.05)
  3-month [Phase II]: number analyzed (Participants) | 19 | 18
  3-month [Phase II] | 3.18 (1.14) | 3.56 (1.00)
  6-month [Phase II]: number analyzed (Participants) | 16 | 16
  6-month [Phase II] | 3.15 (1.10) | 3.77 (.85)

4. Secondary Outcome: Primary Subjective Stressors: Loss of Intimate Exchange
Description: 3-items addressing relationship with relative. Responses include Very much (4), Somewhat (3), Just a little (2), Not at all (1), with higher scores indicating greater loss. Mean of the 3 items is analyzed. Overall mean of participants is reported.
Time Frame: Phase II Baseline, 3-month, 6-month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale (mean)
Arm/Group | Phase II [Randomized]: Treatment | Phase II [Randomized]: Control
Number analyzed (Participants) | 22 | 21
score on a scale (mean)
  Baseline [Phase II] | 3.30 (.92) | 2.86 (.93)
  3-month [Phase II]: number analyzed (Participants) | 19 | 18
  3-month [Phase II] | 3.25 (.97) | 2.98 (.86)
  6-month [Phase II]: number analyzed (Participants) | 16 | 16
  6-month [Phase II] | 3.35 (.82) | 3.13 (.82)

5. Secondary Outcome: Caregiver Distress: Role Captivity
Description: 3-items assessing the involuntary aspects of the caregiving role. Responses for each item include: Very much (4), Somewhat (3), Just a little (2), Not at all (1), with higher score representing greater role captivity. Mean of the 3 items is analyzed. Overall mean of participants is reported.
Time Frame: Phase II Baseline, 3-months, 6-months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale (mean)
Arm/Group | Phase II [Randomized]: Treatment | Phase II [Randomized]: Control
Number analyzed (Participants) | 22 | 21
score on a scale (mean)
  Baseline [Phase II] | 1.97 (.93) | 2.27 (.83)
  3-month [Phase II]: number analyzed (Participants) | 19 | 18
  3-month [Phase II] | 1.98 (1.03) | 2.17 (.77)
  6-month [Phase II]: number analyzed (Participants) | 16 | 16
  6-month [Phase II] | 1.94 (.95) | 2.29 (1.03)

6. Secondary Outcome: Center for Epidemiological Studies Depression (CES-D)
Description: The 20-item Center for Epidemiological Studies Depression (CES-D) survey measure is used to assess respondents' depressive symptoms. Each of the 20 items is scored from 0 = Rarely or none of the time (less than 1 day) to 3 = Most of the time (5-7 days), with 4 items reverse coded. The total CES-D score is summed (ranging 0-60), with higher scores representing more frequent depressive symptoms. Results are reported as a mean of participant scores.
Time Frame: Phase II Baseline, 3-months, 6-months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase II [Randomized]: Treatment | Phase II [Randomized]: Control
Number analyzed (Participants) | 22 | 21
score on a scale
  Baseline [Phase II] | 15.73 (7.11) | 19.10 (7.52)
  3-month [Phase II]: number analyzed (Participants) | 19 | 18
  3-month [Phase II] | 18.47 (8.39) | 21.50 (7.80)
  6-month [Phase II]: number analyzed (Participants) | 16 | 16
  6-month [Phase II] | 18.19 (7.28) | 20.50 (7.21)

7. Other Pre Specified Outcome: Acceptability and Feasibility
Description: This is an author-developed 21-item scale assessing the acceptability and feasibility of the intervention. Response options include Strongly Disagree (1), Disagree (2), Neutral (3), Agree (4), and Strongly Agree (5), or not applicable; 4 items are reverse coded. Higher scores indicate greater acceptability and feasibility of the tool. The summary score represents a mean of the 21-items.
Time Frame: Phase I at 1-month follow up
Population: Phase I [Non-randomized]: All phase I participants completed this set of questions at 1-month.
Measure: Mean (Standard Deviation); unit: score on a scale (mean)
Arm/Group | Phase I [Non-randomized]: Treatment
Number analyzed (Participants) | 20
score on a scale (mean) | 4.22 (0.69)

ADVERSE EVENTS:
Time Frame: Adverse events were documented during study enrollment (following consent through final data collection). Phase I participants did not have any systematic assessment, but were enrolled for a period of about 1 month. A systematic assessment item was implemented during phase II follow up; participants were enrolled for about 6 months.
Description: New or worsening health problems that caused the participant to be unable to perform daily routine (i.e. not go to work or volunteer), seek medical care (i.e. go see your doctor, go to the ER or hospital), or take a new medication
  [Phase I: Non-systematic assessment; Phase II: implemented systematic assessment]
Groups:
- Phase II [Randomized]: Control: Participants randomized to a usual care control group as a part of Phase II.
  Note: If eligible, participants in this control group will be asked if they are interested in enrolling in a similar, additional feature of the study to test the Care to Plan tool following the initial 6-month study.
  Usual Care: Receive care as usual.
  Note: If eligible, participants in this control group will be asked if they are interested in enrolling in a similar, additional feature of the study to test the Care to Plan tool following the initial 6-month study.
Arm/Group | Phase II [Randomized]: Treatment | Phase II [Randomized]: Control | Phase I [Non-randomized]: Treatment
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/22 | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 7/22 | 4/21 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase II [Randomized]: Treatment (N=22) | Phase II [Randomized]: Control (N=21) | Phase I [Non-randomized]: Treatment (N=20)
UTI (Renal and urinary disorders) | 1 | 0 | 0 — Hospitalization related to UTI
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase II [Randomized]: Treatment (N=22) | Phase II [Randomized]: Control (N=21) | Phase I [Non-randomized]: Treatment (N=20)
COVID (Infections and infestations) | 2 | 0 | 0 — Details uncertain [unsure if doctor's visit required]; documented as events for completeness
Initiate Anxiety Medication (Psychiatric disorders) | 1 | 0 | 0
Initiate Thyroid Medication (Endocrine disorders) | 1 | 0 | 0
Hip issue [unspecified] (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Hypertension (Cardiac disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Unknown/not specified medical concern (General disorders) | 0 | 1 | 0 — Staff were not provided details
Eye surgery (Eye disorders) | 1 | 0 | 0 — Uncertain if planned or meets study definition of AE; documented for completeness
Multiple falls during study (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Vulnerable adult report (General disorders) | 1 | 0 | 0 — Filed for caregiver safety and falls; follow up call to APS also made later in study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT03901456/Prot_SAP_000.pdf
  • Informed Consent Form: Phase I (2020-09-29): https://cdn.clinicaltrials.gov/large-docs/56/NCT03901456/ICF_001.pdf
  • Informed Consent Form: Phase II (2021-05-04): https://cdn.clinicaltrials.gov/large-docs/56/NCT03901456/ICF_002.pdf